CLINICAL TRIAL: NCT00618579
Title: A Randomised, Controlled Study Investigating the Safety and Anticoagulant Activity of Administration of Low-molecular-weight Heparin in Healthy Male Subjects Treated With the Monoclonal Anti-factor VIII Antibody, TB-402 and the Safety and Anticoagulant Activity of Administration of TB-402 in Healthy Male Subjects Treated With Warfarin
Brief Title: Effects of LMWH in Healthy Subjects Treated With TB-402 and Effects of TB-402 in Healthy Subjects Treated With Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Collaborators: BioInvent International AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: TB-402-003
Record Dates: First submitted 2008-01-28; First posted 2008-02-20 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Interaction with LMWH or warfarin
MeSH Terms: interventions — TB 402

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LMWH arm - active LMWH (Experimental)
  Interventions: Drug: LWMH in TB-402 treated subjects or TB-402 in warfarin treated subjects
- LMWH arm - placebo (Placebo Comparator)
  Interventions: Drug: LWMH in TB-402 treated subjects or TB-402 in warfarin treated subjects
- Warfarin arm - active warfarin (Experimental)
  Interventions: Drug: LWMH in TB-402 treated subjects or TB-402 in warfarin treated subjects
- Warfarin arm - control (Other)
  Interventions: Drug: LWMH in TB-402 treated subjects or TB-402 in warfarin treated subjects

INTERVENTIONS:
Drug: LWMH in TB-402 treated subjects or TB-402 in warfarin treated subjects — Administration of LMWH in healthy male subjects treated with TB-402 and administration of TB-402 in healthy male subjects treated with warfarin

SUMMARY:
Administration of LMWH in healthy male subjects treated with TB-402 and administration of TB-402 in healthy male subjects treated with warfarin

ELIGIBILITY:
Inclusion Criteria include:

* Males 18 to 45 years of age
* Healthy according to medical history, physical exam, ECG, blood pressure and heart rate, and laboratory profile of blood and urine

Exclusion Criteria include:

* Self or family history of cardiovascular or pulmonary disorder, or coagulation or bleeding disorders or reasonable suspicion of vascular malformations e.g. cerebral haemorrhage, aneurysm or premature stroke
* History of important bleeding episodes
* Previous allergic reaction to immunoglobulin
* Present or previous history of severe allergy, for example asthma or anaphylactic reactions
* FVIII:C <50% at screening
* Clinically significant out of range values for any coagulation test during screening
* Received prescribed medication, over the counter medication or herbal medicines within 14 days of receipt of TB-402

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Anticoagulant activity assessed by aPTT, PT, TGAs and FVIII:c | To study end

SECONDARY OUTCOMES:
Changes in safety parameters over time, PK parameters estimated by NCA, effect of LMWH in TB-402 treated subjects assessed by anti factor Xa (LMWH arm) | To study end

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Jensen, MD, PhD, Principal Investigator — Cyncron CRU
Locations (1):
- Cyncron CRU, Copenhagen, Denmark